CLINICAL TRIAL: NCT00954525
Title: Phase I, Open Label, Dose Escalating Study of Intravenous Ascorbic Acid in Combination With Gemcitabine and Erlotinib in the Treatment of Metastatic Pancreatic Cancer
Brief Title: Intravenous Vitamin C in Combination With Standard Chemotherapy for Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09D.99; JT 1473 (Other: JeffTrial Number)
Record Dates: First submitted 2009-08-04; First posted 2009-08-07 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravenous Vitamin C (Experimental)
  Interventions: Drug: Gemcitabine and Erlotinib; Dietary Supplement: Intravenous Vitamin C

INTERVENTIONS:
Drug: Gemcitabine and Erlotinib — Gemcitabine (dose according to study protocol), Erlotinib (100 mg/day)
Dietary Supplement: Intravenous Vitamin C — 50 grams, 75 grams, or 100 grams of intravenous vitamin C, three times per week for 8 weeks.

SUMMARY:
Eligible candidates will be adults with metastatic pancreatic cancer (confirmed diagnosis with pathology reports and measurable computed tomography (CT) or magnetic resonance imaging (MRI)). Participants must not be receiving any other concurrent chemotherapy, or radiation therapy. Full inclusion/exclusion criteria are available. History and physical examination, and laboratory and imaging analyses will be done within 14 days prior to registration. The three cohorts of subjects will receive 50, 75 or 100 grams of intravenous ascorbic acid, three times per week for 8 weeks. Subjects will also have co-administration of the chemotherapy medications, gemcitabine (intravenously) and erlotinib (orally). Approximately 9 to 18 participants will be enrolled in this Phase I study.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic pancreatic cancer
* Glucose 6 phosphate dehydrogenase status normal
* ECOG performance status 0-2
* Normal creatinine and transaminase
* Women of child-bearing potential confirm negative pregnancy test

Exclusion Criteria:

* Concurrent chemotherapy or radiotherapy
* Significant co-morbid disorders
* Significant psychiatric symptoms
* Prior treatment with gemcitabine
* Concurrent chronic use of immunosuppressive agents (methotrexate, cyclosporine,corticosteroids)
* Regular use of nonsteroidal anti-inflammatory agents
* Smoking more than 1 pack per day
* Excessive alcohol or drug use
* Enrollment in other experimental therapy
* Active infection
* Patients experiencing ongoing response to recent treatments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety, assessed by toxicity (graded by NCI CTC), urinalysis, ECG, basic metabolic panel, CBC, and osmolality. | 8 weeks

SECONDARY OUTCOMES:
Progression-free survival | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Monti, MD, MBA, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Jefferson-Myrna Brind Center of Integrative Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Monti DA, Mitchell E, Bazzan AJ, Littman S, Zabrecky G, Yeo CJ, Pillai MV, Newberg AB, Deshmukh S, Levine M. Phase I evaluation of intravenous ascorbic acid in combination with gemcitabine and erlotinib in patients with metastatic pancreatic cancer. PLoS One. 2012;7(1):e29794. doi: 10.1371/journal.pone.0029794. Epub 2012 Jan 17. PMID 22272248
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/